CLINICAL TRIAL: NCT03992209
Title: Reducing Intraoperative ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter Spp.) Transmission In the Pediatric Operating Room Via Use of a Personal Hand Hygiene System Optimized by OR PathTrac
Brief Title: Reducing Intraoperative Infection Transmission in the Pediatric Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-0759
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Health Care Associated Infection; Hand Hygiene
MeSH Terms: conditions — Cross Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two study arms to include:
  1. Standard hand washing by anesthesia provider
  2. Protocolized hand washing by anesthesia provider
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard handwashing by anesthesia provider (Other): Anesthesia provider will conduct patient care per their usual standard practice in the operating room.
  Interventions: Other: Standard care
- Protocolized hand washing by anesthesia provider (Active Comparator): Anesthesia provider will conduct patient care using a personal hand washing device to optimize hand washing and captures hand washing events in real time.
  Interventions: Other: Protocolized care

INTERVENTIONS:
Other: Standard care — Usual operating room practice
  Arms: Standard handwashing by anesthesia provider
Other: Protocolized care — Hand washing per protocol
  Arms: Protocolized hand washing by anesthesia provider

SUMMARY:
Patients becoming infected during hospitalization occurs frequently and causes harm. It is important for healthcare facilities to take action to prevent these infections and their spread between patients. Despite the presumption of a "sterile" environment, one place where spread of infection is known to happen is in the operating room. This occurs as a result of frequent interaction among healthcare providers, the patient and the environment of the room. Hand washing is an important component of preventing the spread of infections. Scientific evidence has shown that making it easier for people to wash their hands can have two important impacts: (1) reduction of environmental bacterial contamination and (2) reduction in spread of bacterial pathogens. OR PathTrac is new technology that allows tracking of bacterial spread. While data exists about bacterial contamination and transmission in the adult operating room, there is very minimal data about this in the pediatric operating room. Primary aim: To use OR PathTrac to evaluate the effect of a personal hand washing device in reducing operating room exposure to bacterial pathogens in pediatric patients. We hypothesize that this hand washing system will decrease exposure to pathologic bacteria in the pediatric operating room. Secondary aim: To gain knowledge about baseline bacterial contamination and transmission in pediatric operating rooms. We will answer this question by comparing bacterial cultures taken from operating rooms whose personnel are trained to use the hand washing device to operating rooms who are not trained to use the device.

DETAILED DESCRIPTION:
I. Hypotheses: The investigators hypothesize that the use of a personal hand hygiene system by anesthesia providers in the OR, combined with a novel infectious pathogen tracking system will decrease patient exposure to pathologic bacteria in the pediatric operating room.

Primary aim: To use a novel pathogen tracking system (OR PathTrac) to evaluate the effect of a personal hand hygiene device in reducing operating room exposure to bacterial pathogens in pediatric patients.

Secondary aim: To gain knowledge about the baseline bacterial contamination and transmission patterns in pediatric operating rooms.

II. Background and Significance:

Healthcare-associated infections (HAIs) occur frequently and are associated with patient harm. These infections are becoming more difficult to treat due to antibiotic resistance. It is important that healthcare facilities take the necessary steps to prevent the spread of resistant bacteria between patients. ESKAPE bacteria (Enterococcus, S. aureus , Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) are particularly problematic because they have a unique capacity to acquire resistance traits.8 Isolation of these organisms from intraoperative reservoirs has been associated with postoperative infection development.

Many provider-environment-patient interactions occur during routine care in the operating room and must be considered in the development of a successful infection control program. Peaks in environmental contamination that exceed 100 CFU, a threshold associated with high-risk bacterial transmission events repeatedly associated with increased patient mortality and infection, 15 occur during induction and emergence of anesthesia. In turn, these high task density periods correlate with nadirs in hand hygiene (HH) compliance (1.8% HH compliance during induction with 147 environmental CFU and 2.3% HH compliance during emergence with 103 environmental CFU). This work led us to hypothesize that an important consideration for improved OR HH was proximity to the provider.

An intraoperative HH improvement strategy leveraged proximity to the provider and increased provider HH rates 27-fold as compared to those achieved with conventional wall-mounted devices (P < 0.002; 95% confidence interval, 3.3-13.4). Increased HH reduced environmental contamination below 100 CFU (78 fewer colonies per surface sampled; P =0.01). In turn, high risk bacterial transmission events were decreased (32.8% control vs. 7.5% treatment, OR, 0.17; P <0.01), and postoperative HAIs [3.8% treatment vs. 17.2% control, OR 0.19, 95% CI 0.00-0.81, P=0.02, NNT 5.7, including bloodstream, respiratory, urinary tract, and surgical site infections] were reduced.

Much of the aforementioned data has been established in adult operating room patients, there is very little knowledge about this as it pertains to the pediatric operating room. The investigators plan to use a similar evidence-based, hand hygiene improvement strategy to reduce intraoperative transmission of ESKAPE pathogens in the pediatric operating room. After watching a 20-minute instructional video discussing the importance adhering to the many hand hygiene opportunities in the operating room, anesthesia providers will be given a personal hand hygiene device with actionable real-time performance feedback containing 64% ethyl alcohol. The personalized device will be affixed to the provider's waist and will remain there for use throughout the entire case. The number of personal hand hygiene events and a personal hourly hand hygiene rate is visible to the individual providing performance feedback in real time. Devices will be handed out for the case and retrieved on case completion.

The investigators will utilize OR PathTrac, a systematic reservoir collection and software analysis platform, to examine the impact of the device on ESKAPE pathogens. The OR PathTrac system will provide the platform for acquisition of ESKAPE isolates from key reservoirs in the operating room. Systematic phenotypic analysis guided by OR PathTrac will identify epidemiologically related isolates. Related isolates are defined by previously reported thresholds, 12 aligned by temporal association (the reservoir order of collection over time), and mapped to identify bacterial source(s) of transmission. Source identification provides a feedback loop that can be used for proactive optimization of infection control measures. For example, anesthesia resident physician hands are proven to be a typical source of transmission for desiccation tolerant S. aureus isolates that are linked to infection. In the future, this evidence can then be used to proactively optimize the hand hygiene improvement strategy through individual and group level feedback. The OR PathTrac software platform can subsequently measure and report the effectiveness (fidelity) of the improvements, allowing for proactive optimization to achieve sustainability.

III. Research Methods

A. Outcome Measure(s):

Primary outcome measure: The primary endpoint of this study will be the incidence of OR ESKAPE exposure/S. aureus ERTEs with and without the hand hygiene intervention in the pediatric OR.

Secondary outcome measure: Detection and mapping of intraoperative ESKAPE exposure as it pertains to the pediatric operating room.

B. Description of Population to be Enrolled:

This study will include anesthesia providers and pediatric patients, age 1-18 years old, presenting to the main operating room at Children's Hospital Colorado. All, anesthesia providers at Children's Hospital Colorado will be eligible. Patients requiring general anesthesia and placement of a peripheral intravenous catheter will be enrolled.

C. Study Design and Research Methods

Two patients (case pair) undergoing general anesthesia in a randomly selected operating room will be evaluated in a serial manner in order to detect transmission of pathogenic bacteria. A total of 20 case pairs (or 40 patients) will be enrolled. Ten of the case pairs will serve as the intervention group in which the anesthesia provider will be given a personal hand hygiene device to track hand hygiene in real-time. The remaining 10 case pairs will serve as a control group for whom the anesthesia providers will proceed with care per usual practice. Patient care will not change due to their participation in this study, and they will undergo general anesthesia and surgery according to usual practice. Patients will not be asked to perform any tasks for the purpose of the study. The following information will be recorded on the day of surgery:

1. Patients name, case log ID, medical record number. These will be maintained by the research team for approximately 30 days after surgery.
2. Date of surgery, whether it is 1st case vs. 2nd case.
3. Patient diagnosis, ASA (American Society of Anesthesiologists) physical health classification status, age, comorbidities, surgery type & duration, anesthesia provided and duration of anesthesia.
4. Attending Anesthesiologist name with patient case ID log.
5. Wound classification
6. Admitted from (location i.e.: home, unit, etc)

Microbiology cultures will be obtained from three intraoperative reservoirs (patient, anesthesia provider, anesthesia workspace) for each case. Anesthesia induction will occur prior to obtaining patient cultures. A sterile nasal swab will be inserted gently into the internal surface of each nostril & rotated 10 times to culture. In addition, a sterile swab will be inserted gently into the axilla (armpit) and groin of each patient bilaterally & rotated 10 times to culture.

Cultures of the anesthesia provider's hands will be done prior to the case beginning, at the end of the case, and any time they return to the operating room. To collect samples for culture, the provider will be asked to dip their dominant hand into a bag containing sterile sampling solution for 60 seconds. All intraoperative anesthesia providers will potentially be involved. Only those providers who agree to participate will have a culture collected.

Three cultures from the anesthesia workspace (2 from the anesthesia machine and one from the patient's intravenous catheter tubing) will be cultured.

1. APL Valve and Agent Dial Culture

   For case 1-prior to anesthesia care provider entering the OR, 2 sites on the anesthesia machine (adjustable pressure limiting (APL) valve complex & agent dial) will be decontaminated & cultured aseptically. A repeat culture will be obtained at the end of the case. For Case 2, the APL valve and agent dial will not be decontaminated but will be cultured as in case 1.
2. IV Stopcock Culture

Sterile intravenous stopcock sets will be provided preoperatively for each case. The internal lumens of the stopcocks will be cultured on case completion. Microbiology cultures will be obtained by the research team on the day of surgery for each case 1 & case 2. Each culture will be given a study ID & transported to the RDB Bioinformatics laboratory (RDB Bioinformatics, University of Iowa Bioventures Center, 2500 Cross Park Rd, E133, Coralville, IA 52241) at the end of the day using IATA shipping protocols for microbiology assay. No patient or anesthesia care provider information will accompany the samples, and no culture results will be conveyed to the study team. This will ensure that no culture results for a specific person will be known by any study team member. A total of 13 cultures will be obtained from each case for a total of 520 cultures for this study.

D. Description, Risks and Justification of Procedures and Data Collection Tools:

This study presents no more than minimal risk to the participants.

Data Collection Tools:

* Reservoir sampling: OR PathTrac (RDB Bioinformatics, Omaha, NE 68154) collection kits will be used to sample 13 proven reservoirs in each operating room observational unit that is randomly selected for analysis. Reservoirs sampled will include the adjustable pressure-limiting valve and agent dial of the anesthesia machine at case start and at case end (N=2), anesthesia attending physician and primary assigned assistant (resident physician or certified-registered nurse anesthetist) hands before case start and at case end (N=4), the patient nares (both sides), axilla (armpit, both sides), and groin (both sides) after induction and stabilization and at case end prior to emergence (N=6), and the surface of the closed, disinfectable stopcock and/or internal lumen of the open lumen (N=1).
* Demographics: OR number, date, patient age, sex, American Society of Anesthesia (ASA) physical health classification status (I-IV), anesthesia duration (hours), procedure duration (hours), total case duration (hours), comorbidities, preoperative location (same day admit, hospital floor, intensive care unit, other), preadmission yes/no, duration of preadmission (hours), discharge location (post anesthesia care unit, hospital floor, same day unit, intensive care unit, other), dirty or infected surgery yes/no, type of surgery (general abdominal, thoracic, cardiac, general breast, plastics, gynecology/oncology, vascular, etc.), prophylactic antibiotic (yes/no), type of antibiotic and dose, preoperative nasal decolonization (yes/no), type decolonization (povidone iodine, mupirocin, other), days of decolonization, preoperative chlorhexidine (yes/no), concentration and days of chlorhexidine, intraoperative mean and median temperature, postoperative glucose (or other) in mg/dL if measured, surgical provider (assign a code for de-identification), anesthesia provider(s) with de-identified code, postoperative unit location (e.g. 3120 west unit), and same day unit location (e.g. same day room 31).
* Postoperative (within 30 days) elevated white blood cell count yes/no, fever (>38.4 degrees Celsius yes/no), office documentation of infection (yes/no), anti-infective order yes/no, culture positive yes/no, type of culture (sputum, wound, blood, urine, other body fluid). This information will be obtained by chart review by the assistant before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. All intraoperative providers at Children's Hospital Colorado will be eligible to participate
2. Pediatric patients age 1-18 years old presenting to the main operating room at Children's Hospital Colorado who will require general anesthesia with placement of a peripheral intravenous catheter.

Exclusion Criteria:

1. Adult patients, age greater than 18 years old
2. Patients without an intravenous catheter

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Transmission of pathologic bacteria in the operating room | 6 months
  We will use a novel bioinformatics system to track pathogen transmission in the operating room between anesthesia providers, the anesthesia environment and patients.

SECONDARY OUTCOMES:
Baseline pathogen contamination among pediatric surgical patients | 6 months
  We will use culture data to establish what baseline pathogens are present among pediatric operative patients

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Fernandez, MD, Principal Investigator — University of Colorado Department of Anesthesiology
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel TR, Dombrovskiy VY, Lowry SF. Impact of infectious complications after elective surgery on hospital readmission and late deaths in the U.S. Medicare population. Surg Infect (Larchmt). 2012 Oct;13(5):307-11. doi: 10.1089/sur.2012.116. Epub 2012 Oct 19. PMID 23082877
- [Background] Awad SS. Adherence to surgical care improvement project measures and post-operative surgical site infections. Surg Infect (Larchmt). 2012 Aug;13(4):234-7. doi: 10.1089/sur.2012.131. Epub 2012 Aug 22. PMID 22913334
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Magill SS, O'Leary E, Janelle SJ, Thompson DL, Dumyati G, Nadle J, Wilson LE, Kainer MA, Lynfield R, Greissman S, Ray SM, Beldavs Z, Gross C, Bamberg W, Sievers M, Concannon C, Buhr N, Warnke L, Maloney M, Ocampo V, Brooks J, Oyewumi T, Sharmin S, Richards K, Rainbow J, Samper M, Hancock EB, Leaptrot D, Scalise E, Badrun F, Phelps R, Edwards JR; Emerging Infections Program Hospital Prevalence Survey Team. Changes in Prevalence of Health Care-Associated Infections in U.S. Hospitals. N Engl J Med. 2018 Nov 1;379(18):1732-1744. doi: 10.1056/NEJMoa1801550. PMID 30380384
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The epidemiology of Staphylococcus aureus transmission in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):807-18. doi: 10.1213/ANE.0b013e3182a8c16a. PMID 24937345
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Loftus RW, Dexter F, Robinson ADM, Horswill AR. Desiccation tolerance is associated with Staphylococcus aureus hypertransmissibility, resistance and infection development in the operating room. J Hosp Infect. 2018 Nov;100(3):299-308. doi: 10.1016/j.jhin.2018.06.020. Epub 2018 Jun 30. PMID 29966756
- [Background] von Eiff C, Becker K, Machka K, Stammer H, Peters G. Nasal carriage as a source of Staphylococcus aureus bacteremia. Study Group. N Engl J Med. 2001 Jan 4;344(1):11-6. doi: 10.1056/NEJM200101043440102. PMID 11136954
- [Background] Hadder B, Patel HM, Loftus RW. Dynamics of intraoperative Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter transmission. Am J Infect Control. 2018 May;46(5):526-532. doi: 10.1016/j.ajic.2017.10.018. Epub 2018 Feb 12. PMID 29395508
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Background] Rowlands J, Yeager MP, Beach M, Patel HM, Huysman BC, Loftus RW. Video observation to map hand contact and bacterial transmission in operating rooms. Am J Infect Control. 2014 Jul;42(7):698-701. doi: 10.1016/j.ajic.2014.02.021. PMID 24969122
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Loftus RW, Muffly MK, Brown JR, Beach ML, Koff MD, Corwin HL, Surgenor SD, Kirkland KB, Yeager MP. Hand contamination of anesthesia providers is an important risk factor for intraoperative bacterial transmission. Anesth Analg. 2011 Jan;112(1):98-105. doi: 10.1213/ANE.0b013e3181e7ce18. Epub 2010 Aug 4. PMID 20686007
- [Background] Loftus RW, Brown JR, Koff MD, Reddy S, Heard SO, Patel HM, Fernandez PG, Beach ML, Corwin HL, Jensen JT, Kispert D, Huysman B, Dodds TM, Ruoff KL, Yeager MP. Multiple reservoirs contribute to intraoperative bacterial transmission. Anesth Analg. 2012 Jun;114(6):1236-48. doi: 10.1213/ANE.0b013e31824970a2. Epub 2012 Mar 30. PMID 22467892
- [Background] Loftus RW, Patel HM, Huysman BC, Kispert DP, Koff MD, Gallagher JD, Jensen JT, Rowlands J, Reddy S, Dodds TM, Yeager MP, Ruoff KL, Surgenor SD, Brown JR. Prevention of intravenous bacterial injection from health care provider hands: the importance of catheter design and handling. Anesth Analg. 2012 Nov;115(5):1109-19. doi: 10.1213/ANE.0b013e31826a1016. Epub 2012 Oct 9. PMID 23051883
- [Background] Loftus RW, Brindeiro BS, Kispert DP, Patel HM, Koff MD, Jensen JT, Dodds TM, Yeager MP, Ruoff KL, Gallagher JD, Beach ML, Brown JR. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a passive catheter care system. Anesth Analg. 2012 Dec;115(6):1315-23. doi: 10.1213/ANE.0b013e31826d2aa4. Epub 2012 Nov 9. PMID 23144441
- [Background] Clark C, Taenzer A, Charette K, Whitty M. Decreasing contamination of the anesthesia environment. Am J Infect Control. 2014 Nov;42(11):1223-5. doi: 10.1016/j.ajic.2014.07.016. Epub 2014 Oct 30. PMID 25444268
- [Background] Dancer SJ, Stewart M, Coulombe C, Gregori A, Virdi M. Surgical site infections linked to contaminated surgical instruments. J Hosp Infect. 2012 Aug;81(4):231-8. doi: 10.1016/j.jhin.2012.04.023. Epub 2012 Jun 15. PMID 22704634
- [Derived] Fernandez PG, Dexter F, Brown J, Whitney G, Koff MD, Cao S, Loftus RW. Epidemiology of Enterococcus , Staphylococcus aureus , Klebsiella , Acinetobacter , Pseudomonas , and Enterobacter Species Transmission in the Pediatric Anesthesia Work Area Environment With and Without Practitioner Use of a Personalized Body-Worn Alcohol Dispenser. Anesth Analg. 2024 Jan 1;138(1):152-160. doi: 10.1213/ANE.0000000000006326. Epub 2023 Dec 14. PMID 36623234